CLINICAL TRIAL: NCT06369545
Title: Examination of the Efficacy of ESWT (Extracorporeal Shock Wave Therapy) and TENS (Transcutaneous Electrical Nerve Stimulation) in Individuals Receiving Drug Treatment for Chronic Pelvic Pain Syndrome: Randomized Controlled Study
Brief Title: Chronic Pelvic Pain Syndrome in Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Ugur Cavlak, Clinical Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BiruniUniver
Record Dates: First submitted 2024-03-29; First posted 2024-04-17 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Pelvic Pain Syndrome
Keywords: Chronic Pelvic Pain Syndrome; Male; ESWT; TENS
MeSH Terms: interventions — Exercise; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized Controled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP I: TENS (Experimental): PHYSIOTHERAPY PROGRAM PLUS TENS
  Interventions: Other: EXERCISE; Other: TENS
- GROUP II: ESWT (Active Comparator): PHYSIOTHERAPY PROGRAM PLUS ESWT
  Interventions: Other: EXERCISE; Other: ESWT

INTERVENTIONS:
Other: EXERCISE — All participants included in this group will receive Exercises
Other: TENS — All participants included in this group will receive TENS
  Arms: GROUP I: TENS
Other: ESWT — All participants included in this group will receive ESWT
  Arms: GROUP II: ESWT

SUMMARY:
The aim of this study is to evaluate the effectiveness of ESWT (Extracorporeal Shock Wave Therapy) and TENS (Transcutaneous Electrical Nerve Stimulation) in individuals diagnosed with chronic pelvic pain syndrome and treated with medication. The study was organized as a randomized controlled trial. The sample size is 30 patients suffering from chronic pelvic pain syndrome.

DETAILED DESCRIPTION:
Volunteers who are between the ages of 20-40, diagnosed with chronic pelvic pain syndrome, and who meet the inclusion criteria will be included in the study and will be randomized into 2 groups: Group I (TENS) and Group II (ESWT).

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 20-40 years old males
2. Diagnosis of Chronic Pelvic Pain Syndrome

Exclusion Criteria:

1. Cancer
2. Surgery related to pelvic floor

2. Receiving drug treatment

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
VISUAL ANALOUGE SCALE | baseline and immediately after the intervention
  It evaluates pain intensity grading between 0-10. Higher score shows severe pain.
National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) | baseline and immediately after the intervention
  This assesses the quality of life. The index has sub dimensions(pain, urinary symptoms, quality of life impact).
  The score evaluation of the pain scale is between 1 and 21 points, the score evaluation of the urination scale is between 0 and 10 points, and the score evaluation of the quality of life scale is between 0 and 12 points.
ALGOMETER | baseline and immediately after the intervention
  This evaluates pain tolerance threshold of the patients.The less score shows pain intolerance.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale- HAD | baseline and immediately after the intervention
  This evaluates depresive symtoms of the patients.This scale is a self-rating scale. The scale is a 4-point Likert type scale consisting of 14 items in total, including anxiety and depression subscales (Aydemir, Güvenir, Küey, & Kültür, 1997). 7 items in the scale are for anxiety and 7 items are for depression. Participants will be asked to mark each item considering the situation they have experienced in the last week. Each item contains four options. Options will be scored between 0-3 points. The lowest score for the anxiety and depression subscales is 0 and the highest score is 21 points.
Nottingham Health Profile-NHP | baseline and immediately after the intervention
  This evaluates quality of life of the patients. The survey consists of 6 sections. These sections are pain, emotional reactions, social isolation, physical activity, energy and sleep. It consists of 38 items in total. Each section is scored between 0-100 points. 0 will be considered the best score and 100 will be considered the worst score.
Digital Muscle Testing | baseline and immediately after the intervention
  To evaluate muscles's strenght using by Power Track. Higher cosre shows good strneght.
Flexibility Measurements | baseline and immediately after the intervention
  To measure flexibility of the muscles, manually. The amount of elasticity is measured and the result is recorded in cm.
ROM Assessments | baseline and immediately after the intervention
  To measure range of motion of the joints by using goniometer.
Lasegue Test | baseline and immediately after the intervention
  To measure flexibility of the sciatic nerve, manually.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences in Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schneider MP, Tellenbach M, Mordasini L, Thalmann GN, Kessler TM. Refractory chronic pelvic pain syndrome in men: can transcutaneous electrical nerve stimulation help? BJU Int. 2013 Jul;112(2):E159-63. doi: 10.1111/bju.12005. Epub 2013 Feb 22. PMID 23433012